CLINICAL TRIAL: NCT05269888
Title: An Observational Study to Evaluate Immune Response to Covid-19 Vaccines, Infections and Immune Treatments in People With Multiple Sclerosis
Brief Title: Covid-19 Vaccine Immune Response in Multiple Sclerosis
Acronym: CoVaR-MS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3200
Record Dates: First submitted 2022-03-02; First posted 2022-03-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Study group - Ocrelizumab: 30 patients with multiple sclerosis on Ocrelizumab (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - Natalizumab: 30 patients with multiple sclerosis on Natalizumab (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - Alemtuzumab: 30 patients with multiple sclerosis on Alemtuzumab (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - Tecfidera: 30 patients with multiple sclerosis on Tecfidera (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - Fingolimod: 30 patients with multiple sclerosis on Fingolimod (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - Interferon: 30 patients with multiple sclerosis on Interferon (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Study group - off DMT: 30 patients with multiple sclerosis off disease modification treatment (DMT) (standard of care)
  Interventions: Other: Blood Test 1; Other: Blood Test 2
- Control group: 30 healthy volunteers
  Interventions: Other: Blood Test 1; Other: Blood Test 2

INTERVENTIONS:
Other: Blood Test 1 — Blood test 1 - At 12 months (+3months) from the date of 1st Covid-19 vaccine:
  Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche, T-SPOT® COVID SARS-CoV-2, Full Blood Count, Serum Immunoglobulins, Anti-VZV titres
Other: Blood Test 2 — Blood test 2 - At 18 months (+3months) from the date of 1st Covid-19 vaccine:
  Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche, T-SPOT® COVID SARS-CoV-2, Full Blood Count, Serum Immunoglobulins, Anti-VZV titres

SUMMARY:
Coronavirus (Covid-19) has affected millions of people worldwide. Vaccines to prevent Covid-19 infection have been offered to reduce the risk of infection. While these vaccines have been offered to people with multiple sclerosis (MS), they have not been tested in these individuals. It is uncertain whether people with MS will develop protective antibodies after a Covid-19 vaccination and how long these antibodies will last.

The investigators are planning to study the immune response to the full course of Covid-19 vaccine in people with MS (study group) and compare this to people without MS or immune suppression (control group).

ELIGIBILITY:
Inclusion Criteria (Study Group - MS Patients):

* Aged 18 years and over
* Diagnosis of Multiple Sclerosis as per McDonald's Criteria 2017
* Falls into one of following the Disease Modification Treatment (DMT) groups: on Ocrelizumab, on Natalizumab, on Alemtuzumab, on Tecfidera, on Fingolimod, on Interferon, not on any DMT
* Has had a complete course of Covid-19 vaccination including any boosters (standard dosing: prescribed as per the UK Government guidelines)
* Willing and able to give fully informed consent
* Willing and able to comply with the study procedures

Exclusion Criteria (Study Group - MS Patients):

* Has declined or does not wish to have Covid-19 vaccine
* Has switched DMT since the date of first dose of Covid-19 vaccine
* Has any other immunological condition or on immune treatment causing immune suppression
* Has declined or does not wish to have Covid-19 vaccine
* Ineligible* for Covid-19 vaccine (*Ineligible for health reasons and/or as per Government prioritisation of vaccinations)
* Non-English speaker where translation facilities are insufficient to guarantee informed consent

Inclusion Criteria (Control Group - Healthy Volunteers):

* Aged 18 years and over
* Has had a complete course of Covid-19 vaccination (standard dosing: prescribed as per the UK Government guidelines)
* Willing and able to give fully informed consent
* Willing and able to comply with the study procedures

Exclusion Criteria (Control Group - Healthy Volunteers):

* Has declined or does not wish to have Covid-19 vaccine
* Has MS or another long-term immunological condition
* History of taking any immune treatment causing immune suppression in the last 5 years
* History of any immune conditions or comorbidities known to result in immune suppression within the last 5 years;
* Ineligible* for Covid-19 vaccine (*Ineligible for health reasons and/or as per Government prioritisation of vaccinations)
* Currently participating in one or more interventional trials involving immune suppression or immune agent
* Non-English speaker where translation facilities are insufficient to guarantee informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are two groups of participants in this study:
  1. Multiple Sclerosis Patients (Study Group): 210 patients with multiple sclerosis, on and off disease modification treatment (DMT):
     * 180 patients on DMT, divided as follows: 30 patients on Ocrelizumab, 30 patients on Natalizumab, 30 patients on Alemtuzumab, 30 patients on Tecfidera, 30 patients on Fingolimod, 30 patients on Interferon
     * 30 patients off DMT
  2. Healthy Volunteers (Control Group): 30 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood titres of Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche in MS patients compared with healthy volunteers 12 months from date of first dose of Covid-19 vaccine | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche
Blood titres of Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche in MS patients compared with healthy volunteers 18 months from date of first dose of Covid-19 vaccine | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Anti-SARS-CoV-2 S1/S2/N IgG antibody Roche
T-SPOT® COVID SARS-CoV-2 test status in MS patients compared with healthy volunteers 12 months from date of first dose of Covid-19 vaccine | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  T-SPOT® COVID SARS-CoV-2 test status
T-SPOT® COVID SARS-CoV-2 test status in MS patients compared with healthy volunteers 18 months from date of first dose of Covid-19 vaccine | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  T-SPOT® COVID SARS-CoV-2 test status

SECONDARY OUTCOMES:
Type and timing of DMT in MS patients | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Type and timing of DMT
Type and timing of DMT in MS patients | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Type and timing of DMT
Type and timing of Covid-19 vaccine in MS patients compared with healthy volunteers | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Type and timing of Covid-19 vaccine
Type and timing of Covid-19 vaccine in MS patients compared with healthy volunteers | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Type and timing of Covid-19 vaccine
Participant-reported PCR positive Covid-19 infection/s in MS patients compared with healthy volunteers | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Participant-reported PCR positive Covid-19 infection/s
Participant-reported PCR positive Covid-19 infection/s in MS patients compared with healthy volunteers | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Participant-reported PCR positive Covid-19 infection/s
Covid-19 vaccine-related serious adverse events in MS patients compared with healthy volunteers | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Vaccine-related serious adverse events
Covid-19 vaccine-related serious adverse events in MS patients compared with healthy volunteers | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Vaccine-related serious adverse events
Demographics of MS patients compared with healthy volunteers | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Demographics
Demographics of MS patients compared with healthy volunteers | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Demographics
Co-morbidity status of MS patients compared with healthy volunteers | 12 months (+3 months) from date of first dose of Covid-19 vaccine
  Co-morbidity status
Co-morbidity status of MS patients compared with healthy volunteers | 18 months (+3 months) from date of first dose of Covid-19 vaccine
  Co-morbidity status

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom